CLINICAL TRIAL: NCT02160093
Title: Impact of Chronic Disease Control and Aging Psychology on Outcomes of Frailty-Sarcopenia Syndrome in Ambulatory Geriatric Patients
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201404030RIND
Record Dates: First submitted 2014-06-03; First posted 2014-06-10 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Ambulatory Geriatric Outpatients at High Risk of Frailty
Keywords: sarcopenia; frailty; chronic disease control; aging psychology
MeSH Terms: conditions — Sarcopenia; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Pursuant to our previous longitudinal study (ClinicalTrials.gov ID: NCT02073370) in geriatric outpatients cooperated with the Department of Family Medicine, Department of Geriatrics and Gerontology, National Taiwan University Hospital, this study will be conducted to examine the impacts of the specific co-morbidities and ageing psychology on the outcomes of frailty/sarcopenia syndrome. The thresholds of specific chronic disease will be reviewed after frailty being considered in the elderly with co-morbidity condition. In addition, the conceptual framework and corresponding measuring instrument of "mental frailty" will be expected developed.

ELIGIBILITY:
Inclusion criteria : compatible one of following conditions

* functional decline in recent one year
* cognitive function decline
* depressive symptom
* mobility impairment
* fall in recent one year
* eating or feeding problems/weight loss
* co-morbid conditions≧5
* tracking by different physician ≧3 in recent half year
* polypharmacy≧8 in recent 3 months
* hospitalization ≧1 in recent one year
* emergency visits≧2 in recent one year
* aged ≧ 80

Exclusion criteria:

* non-ambulatory (bed-ridden) patients
* long-term residents at nursing homes
* patients with a life expectancy shorter than six months
* impairment in vision, hearing, or communicative ability
* making convenience of clinical evaluation during the study period impossible.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Ambulatory geriatric outpatients aged 65 and over from NTUH
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2014-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Operation instrument of mental frailty for older adults | Up to 2 years
  The psychological adaptation to aging is a dynamic process. The dynamic process and the Selection-Optimization-Compensation process will have their effect on the actual coping actions in everyday life. The instruments will be set up to evaluate the aging psychology process

SECONDARY OUTCOMES:
Compare the well chronic disease control and inappropriate condition on the dynamic frail transitions in ambulatory geriatric outpatients | up to 4 years
  The records of chronic disease control status of the same ambulatory geriatric outpatients from previous study, "Clinical evaluation, biomarkers and metabolomics of sarcopenia in frail older adults at ambulatory clinics", will be linked to this study.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Yu Chen, MD, Principal Investigator — National Taiwan University, College of Medicine
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan